CLINICAL TRIAL: NCT06801171
Title: Randomized Clinical Trial Testing a Mixed Intervention to Improve Resilience in People Aged Over 60 Years With Neurocognitive Disorders.
Brief Title: A Mixed Intervention to Improve Resilience for Patient With Neurocognitive Disorders
Acronym: RESILIENCE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24-AOI-02
Record Dates: First submitted 2025-01-17; First posted 2025-01-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Disorder
Keywords: neurocognitive disorder; resilience; mixed intervention
MeSH Terms: conditions — Cognitive Dysfunction; Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: monocentric interventional study with minimal risks randomized into three parallel groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): group without intervention
- cognitive stimulation (Experimental): group with 12 sessions in group of cognitive stimulation
  Interventions: Other: cognitive stimulation
- mixed intervention (Experimental): group with 12 sessions in group of mixed stimulation (yoga, cognitive behavioral therapy, mindfulness meditation, positive psychology)
  Interventions: Other: mixed intervention

INTERVENTIONS:
Other: cognitive stimulation — 12 sessions (one per week for 12 weeks) in group of cognitive stimulation
  Arms: cognitive stimulation
Other: mixed intervention — 12 sessions (one per week for 12 weeks) in group of mixte stimulation (yoga, cognitive behavioral therapy, mindfullness meditation, positive psychology)
  Arms: mixed intervention

SUMMARY:
The study aims to test a program combining cognitive behavioral therapy techniques, positive psychology techniques, mindfulness meditation and yoga, in order to improve resilience in patient with minor cognitive disorder.

This intervention will be compared to a control group, but also with a group testing another intervention (an intervention that does not improve resilience in the elderly, namely a "cognitive stimulation" intervention) in order to ensure that the effect potentially obtained is not due to the simple management of the participant.

The duration of the intervention will be 3 months, with an evaluation directly before and after the intervention.

In addition, in order to best evaluate the effectiveness of the interventions over time, two follow-up measurements will be proposed: a measurement one month after the intervention, then a final one three months after the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Man or Woman aged > 60 years
2. Have a minor neurocognitive disorder according to the criteria of the DSM 5
3. Score of 145 or less on the Wagnild and Young Resilience Scale (RS) (Wagnild, 2009).
4. Subject able to read and write French;
5. Subject beneficiaries of a social security scheme;
6. Ability to understand and sign free and informed consent.

Exclusion Criteria:

1. Subject already practicing meditation and/or yoga and/or Tai Chi
2. Subject currently undergoing psychological therapy (whatever the approach)
3. Subject with a major hearing, visual or motor disability likely to interfere with the proposed interventions or the performance of assessments;
4. Presence and/or recent history (within the last 5 years prior to inclusion in the study) of major psychiatric disorders (e.g., schizophrenia, severe depression, addiction, bipolar disorders, psychotic disorders, risk of dissociation, panic attack, generalized anxiety disorder, etc.)
5. If taking psychotropic treatment, the dose must have been stable for 4 weeks
6. Vulnerable persons are defined in Articles L1121-5 to -8

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of resilience of patients suffering from mild neurocognitive disorder (NCD) compared to a passive control group (without any intervention). | Pre intervention
  Comparison of scores at Resilience Scale for Older Adults (RSOA) between group control and mixed intervention mixed Questionnaire adapted for older adults to evaluate resilience. The RSOA questionnaire contains 33 questions which consists of four overarching factors and 11 facets. The Intrapersonal factor consists of Perseverance and Determination, Self-Efficacy and Independence, Purpose and Meaning, and Positive Perspective. The Interpersonal factor consists of Sense of Community, Family Support, and Friend/Neighbour Support. The Spiritual factor consists of Faith and Prayer, and the Experiential factor consists of Previous Adversity and Proactivity.
  Each question is measured using a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree) Higher scores indicate a higher resilience.
Improvement of resilience of patients suffering from mild neurocognitive disorder (NCD) compared to a passive control group (without any intervention). | Pre intervention
  Comparison of scores at Resilience Scale (RS) between group control and mixed intervention mixed
  The RS questionnaire contains 25 questions. The items in the resilience scale address different aspects of the ability to cope with difficulties and bounce back. For example, some statements concern the ability to find meaning in stressful situations, to remain hopeful for the future, or to feel supported by those around one.
  Each question is measured using a 5-point Likert scale from 1 (strongly disagree) to 7(strongly agree) Higher scores indicate a higher resilience
Improvement of resilience of patients suffering from mild neurocognitive disorder (NCD) compared to a passive control group (without any intervention). | Pre intervention
  Comparison of scores at Brief-COPE between group control and mixed intervention mixed The Brief-COPE is a self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Coping" is defined broadly as an effort used to minimise distress associated with negative life experiences.
  The questionnaire contains 28 questions. Each question is measured using a 4-point Likert scale from 1 I haven't been doing this at all to 4= I've been doing this a lot Higher scores indicate a better coping.

SECONDARY OUTCOMES:
Persistence of improvement in resilience over time | Through study completion, an average of 3 months
  Comparison of scores at Resilience Scale for Older Adults (RSOA) at different time points The RSOA questionnaire contains 33 questions which consists of four overarching factors and 11 facets. The Intrapersonal factor consists of Perseverance and Determination, Self-Efficacy and Independence, Purpose and Meaning, and Positive Perspective. The Interpersonal factor consists of Sense of Community, Family Support, and Friend/Neighbour Support. The Spiritual factor consists of Faith and Prayer, and the Experiential factor consists of Previous Adversity and Proactivity.
  Each question is measured using a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree)
  Higher scores indicate a higher resilience.
Persistence of improvement in resilience over time | Through study completion, an average of 3 months
  Comparison of scores at Resilience Scale (RS) at different time points The RS questionnaire contains 25 questions. The items in the resilience scale address different aspects of the ability to cope with difficulties and bounce back. For example, some statements concern the ability to find meaning in stressful situations, to remain hopeful for the future, or to feel supported by those around one.
  Each question is measured using a 5-point Likert scale from 1 (strongly disagree) to 7(strongly agree) Higher scores indicate a higher resilience
Persistence of improvement in resilience over time | Through study completion, an average of 3 months
  Comparison of scores at Brief-COPE at different time points The Brief-COPE is a self-report questionnaire designed to measure effective and ineffective ways to cope with a stressful life event. Coping" is defined broadly as an effort used to minimise distress associated with negative life experiences.
  The questionnaire contains 28 questions. Each question is measured using a 4-point Likert scale from 1 I haven't been doing this at all to 4= I've been doing this a lot
  Higher scores indicate a better coping.

CONTACTS AND LOCATIONS:
Overall Officials: SACCO GUILLAUME, Pr, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice
Locations (1):
- CHU de Nice, Nice, France

IPD SHARING:
Plan to Share IPD: No